CLINICAL TRIAL: NCT05674877
Title: Opioid Sparing Anesthesia in Patients With Liver Cirrhosis Undergoing Liver Resection: A Controlled Randomized Double Blind Study
Brief Title: Opioid Sparing Anesthesia in Patients With Liver Cirrhosis Undergoing Liver Resection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed Youssef Ollaek, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 00309/2022
Record Dates: First submitted 2022-12-20; First posted 2023-01-09 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Liver Cirrhosis
Keywords: Dexmedetomidine; ketamine; Liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Sodium Chloride; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid-based group (OB) (Placebo Comparator): .Patients in the opioid-based group will receive placebo boluses and infusions of saline.
  The intra-operative hemodynamics target will be to maintain the mean arterial blood pressure and heart rate within 20% of baseline value. Significant hemodynamic alterations will be managed as follows:
  Hypertension and/or tachycardia defined as more than 20% increase of the baseline readings will be managed by top-up doses of fentanyl 1µg/kg
  Interventions: Drug: Opioid-based group (OB) (placebo/saline)
- Opioid sparing group (OS) (Active Comparator): Patients in the Opioid Sparing group will receive a loading dose of dexmedetomidine (1µg/kg over 10 minutes). This will be followed by a fixed continuous maintenance infusion of 0.5µg/kg/hour. Furthermore, a single induction analgesic dose of 0.5 mg/kg ketamine will be given to all patients in the OS group. This will be followed by 0.25 mg/kg/h continuous maintenance infusion. Dexmedetomidine and ketamine infusions will be stopped 30 minutes prior to the conclusion of surgery.
  The intra-operative hemodynamics target will be to maintain the mean arterial blood pressure and heart rate within 20% of baseline value. Significant hemodynamic alterations will be managed as follows:
  Hypertension and/or tachycardia defined as more than 20% increase of the baseline readings will be managed by top-up doses of fentanyl 1µg/kg in the two study groups.
  Interventions: Drug: Opioid sparing group (OS) (dexmedetomidine (PRECEDEX™ "dexmedetomidine hydrochloride" - Pfizer) and ketamine)

INTERVENTIONS:
Drug: Opioid-based group (OB) (placebo/saline) — Patients in the opioid-based group will receive placebo boluses and infusions of saline.
  Other Names: OB
  Arms: Opioid-based group (OB)
Drug: Opioid sparing group (OS) (dexmedetomidine (PRECEDEX™ "dexmedetomidine hydrochloride" - Pfizer) and ketamine) — Patients in the Opioid Sparing group will receive a dexmedetomidine (PRECEDEX™ "dexmedetomidine hydrochloride" - Pfizer) and ketamine.
  Other Names: OS
  Arms: Opioid sparing group (OS)

SUMMARY:
This randomized clinical trial will investigate the opioid sparing effect of dexmedetomidine and ketmine infusion in cirrhotic patients undergoing liver resection

DETAILED DESCRIPTION:
Patient enrollment will start after approval of the study protocol by the local Ethics and Research Committee and the Institutional Review Board (IRB) of the Departments of Anesthesia, ICU and Pain Management and the National Liver Institute, Faculty of Medicine, Menoufia University. The study will be conducted in the Anesthesia Department, National Liver Institute and will be registered with the ClinicalTrials.gov (http://www.clinicaltrials.gov) before patients enrollment.

The study will include adult patients with liver cirrhosis undergoing liver resection. Patients will be randomly allocated into one of the two study groups using an online randomization program (http://www.randomizer.org). Random allocation numbers will be concealed in opaque closed envelops. A written informed consent will be taken from each patient.

Five leads electrocardiography, pulse oximetry and peripheral perfusion index using masimo pulse oxymetry finger prope (Masimo, Irvine,CA, USA), end-tidal CO2, invasive arterial blood pressure, central venous pressure, The electrical cardiometry (EC) (ICON monitor; Cardiotronics Inc., La Jolla, CA, USA) for cardiac output monitoring (CO). oesophageal temperature, fraction inspired oxygen concentration, fraction inspired and expired desflurane. Bispectral index will be used to monitor the depth of anesthesia (BIS Covidien USA.), The neuromuscular function will be monitored using TOF-Watch SX (Schering-Plough, Swords, Co. Dublin, Ireland).

All patients fulfilling the study inclusion criteria will undergo a thorough clinical evaluation including laboratory assessment of liver and renal functions. Other diagnostic and/or laboratory workup will be requested by the attending anesthetist and the surgeon according to the patient clinical condition and the proposed surgical intervention.

Bilateral transversus abdominis plane (TAP) block:

All patients in the two study groups will receive a single shot ultrasound-guided bilateral TAP block using levopubivacaine. The effectiveness and dermatomal distribution of the block will be checked after 30 minutes and before induction of general anesthesia.

Anesthesia will be induced in all patients using fentanyl 2µg/kg, propofol 2 mg/kg, and rocuronium 0.6 mg/kg to facilitate endotracheal intubation. After induction of anesthesia, patients will be randomly allocated in two groups opioid sparing group (OS) and opioid-based group (OB). Patients in the Opioid Sparing group will receive a loading dose of dexmedetomidine (1µg/kg over 10 minutes). This will be followed by a fixed continuous maintenance infusion of 0.5µg/kg/hour. Furthermore, a single induction analgesic dose of 0.5 mg/kg ketamine will be given to all patients in the OS group. This will be followed by 0.25 mg/kg/h continuous maintenance infusion. Dexmedetomidine and ketamine infusions will be stopped 30 minutes prior to the conclusion of surgery. Patients in the opioid-based group will receive placebo boluses and infusions of saline. The attending anesthesiologist will be blinded to the patient group assignment.

Anesthesia will be maintained with a mixture of air, oxygen and desflurane to keep a BIS between 40 and 60. Muscle relaxation will be maintained by additional top-up doses of rocuronium 0.15mg/kg and will be guided by the response to ulnar nerve stimulation. Ventilation parameters will be adjusted to maintain normocapnia. Intraoperative normothermia will be maintained using a forced air warm blanket (Model 750-Bair Hugger Temperature Management Unit, SMA MISR, Arizant Healthcare Inc, USA), a humidifier, and warm intravenous fluids. Deep venous thrombosis (DVT) prophylaxis will include elastic stockings, sequential compression device (SCD) (Kendall Company, Tyco, USA) on the lower limb until early ambulation. Intraoperative fluid, fresh frozen plasma, and blood replacement therapy will be guided by the continuous monitoring of the central venous pressure and EC Cardiometry. and will be titrated to maintain hemodynamic stability and a hemoglobin level of 10 g/dL.

The intra-operative hemodynamics target will be to maintain the mean arterial blood pressure and heart rate within 20% of baseline value. Significant hemodynamic alterations will be managed as follows:

* Bradycardia (heart rate < 50 beats/min) will be managed by incremental 0.5 mg doses of atropine.
* Hypertension and/or tachycardia defined as more than 20% increase of the baseline readings will be managed by top-up doses of fentanyl 1µg/kg in the two study groups.
* Hypotension defined as more than 20% reduction in the baseline mean arterial blood pressure will be managed by incremental doses of ephedrine 5mg in the two study groups.

At the end of surgery and when two responses to train-of-four ulnar nerve stimulation are detected (T2), residual rocuronium-induced neuromuscular block will be antagonized by sugammadex 2 mg/kg. Patients will be discharged to the surgical intensive care unit after extubation. Postoperative analgesia will be achieved using patient-controlled fentanyl infusion (PCA fentanyl).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with liver cirrhosis [Child A] aged 18 to 65 years undergoing liver resection.
* American Society of Anesthesiologists class II-III.

Exclusion Criteria:

* Renal or cardiac dysfunction
* History of chronic pain
* Alcohol or drug abuse
* Analgesic use in last 24 hours before surgery
* Major intraoperative hemodynamic instability
* The need for postoperative ventilation
* Psychiatric disorders
* Inability to comprehend pain assessment
* Allergy or contraindication to any of the study medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Intraoperative fentanyl requirements | Through operative time
  Intraoperative fentanyl requirements in micrograms

SECONDARY OUTCOMES:
Postoperative PCA fentanyl requirements | Postoperative over 48 hours
  Postoperative patient controlled analgesia (PCA) fentanyl requirements in micrograms
Incidence of severe postoperative opioid related adverse events | 48 hours after extubation
  desaturation episodes (on room air), postoperative nausea and vomiting and postoperative ileus.
  Desaturation is defined as a decrease of oxygen saturation equal to or exceeding 4% of the baseline value.
  Postoperative ileus defined as absence of flatus or stools
Incidence of bradycardia | Through operative time
  heart rate < 50 beats/min
Incidence of hypotension | Through operative time
  Hypotension defined as more than 20% reduction in the baseline mean arterial blood pressure
Incidence of hypertension | Through operative time
  Hypertension defined as more than 20% increase of the baseline readings
Extubation time | Time from antagonist administration till extubation
  Time from antagonist administration till extubation
Postoperative pain score (VAS) score | 2 hours after extubation then every 6 hours for 48 hours
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 (no pain) and 10 (pain as bad as it could possibly be)
ICU and hospital length of stay | Immediate postoperative to maximum of 28 days
  Defined as the number of days after extubation before first hospital discharge
Average required end-tidal desflurane | Through operative time
  meaured in percentage
Surgical time | Through operative time
  From skin incision to closure measured in minutes
Anesthesia time | Through operative time
  From induction to extubation measured in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed C Ollaek, Principal Investigator — Department of Anesthesia, Surgical ICU and Pain Management
Locations (1):
- National Liver Institute, Menoufia University, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: No